CLINICAL TRIAL: NCT04165863
Title: Effectiveness of Treatment With Rich Platelet Fibrin (PRF) VS Gold Standard in the Healing Process of Surgical Wounds in Patients Undergoing Knee Replacement
Brief Title: Effectiveness of Treatment With Rich Platelet Fibrin (PRF) VS Gold Standard in Patients Undergoing Knee Replacement
Acronym: Fibrin4Fast
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Fibrin4Fast
Record Dates: First submitted 2019-11-14; First posted 2019-11-18 (Actual); Last update posted 2022-01-19 (Actual); Status verified 2019-11

CONDITIONS: Knee Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A (Experimental): treatment of the surgical wound healing process with Platelet-rich-fibrin in patients undergoing total knee replacement surgery
  Interventions: Procedure: total knee replacement surgery
- B (Active Comparator): Gold standard treatment of the surgical wound healing process without Platelet-rich-fibrin in patients undergoing total knee replacement surgery
  Interventions: Procedure: total knee replacement surgery

INTERVENTIONS:
Procedure: total knee replacement surgery — total knee replacement surgery

SUMMARY:
Randomized controlled single blind trial for the evaluation of the treatment of the surgical wound healing process with Platelet-Rich-Fibrin compared to the gold standard (without Platelet-Rich-Fibrin) in patients undergoing knee replacement.

ELIGIBILITY:
Inclusion Criteria:

* Males or females undergoing a total knee prosthesis.
* Willingness and ability to comply with the study procedures and visit schedules and ability to follow verbal and written instructions.
* Hb > 11 g/dl; Platelet value > 150.000 plt/mmc;
* Patients with non clinical alteration of ECG;
* Signature of informed consent;

Exclusion Criteria:

* Patients incapable of understanding and of wanting;
* Systemic disorders such as diabetes, rheumatic diseases;
* Patients with malignancy;
* Thyroid metabolic disorders ;
* Abuse of alcohol, drugs and pharmaceutical drugs
* Body mass index > 40;

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2020-01-20 (Actual); Primary Completion 2021-11-04 (Actual); Study Completion 2021-11-04 (Actual)

PRIMARY OUTCOMES:
clinical improvement of the healing process | 2 weeks
  Clinical improvement of the healing process, assessed by application of the Hollander Wound Evaluation Scales at 2 weeks of follow up

SECONDARY OUTCOMES:
Dermatology life quality | 3 days, 15 days and 1 month
  Dermatology life quality index improvement at 3 days, 15 days and 1 month

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Itituto Ortopedico Rizzoli, Bologna, BO, Italy

REFERENCES:
- [Result] Harato K, Tanikawa H, Morishige Y, Kaneda K, Niki Y. What are the important surgical factors affecting the wound healing after primary total knee arthroplasty? J Orthop Surg Res. 2016 Jan 13;11:7. doi: 10.1186/s13018-016-0340-y. PMID 26762213
- [Result] Galat DD, McGovern SC, Larson DR, Harrington JR, Hanssen AD, Clarke HD. Surgical treatment of early wound complications following primary total knee arthroplasty. J Bone Joint Surg Am. 2009 Jan;91(1):48-54. doi: 10.2106/JBJS.G.01371. PMID 19122078
- [Result] Rui M, Zheng X, Sun SS, Li CY, Zhang XC, Guo KJ, Zhao FC, Pang Y. A prospective randomised comparison of 2 skin closure techniques in primary total hip arthroplasty surgery. Hip Int. 2018 Jan;28(1):101-105. doi: 10.5301/hipint.5000534. PMID 29148019